CLINICAL TRIAL: NCT00423176
Title: Efficacy and Safety of 200mcg BID Mometasone Furoate Nasal Spray (MFNS) Versus Placebo as Adjunctive Treatment to Antibiotics in Relief of Symptoms of Acute Bacterial Sinusitis
Brief Title: The Study of Nasonex® Compared With Placebo for the Relief of Symptoms Associated With Acute Bacterial Sinusitis When Used With Antibiotics (Study P04824AM3)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on business priorities. Not related to any safety or efficacy issue & took place before data were unblinded or analyzed
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04824
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2022-02

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MFNS + Antibiotic (Experimental): Mometasone furoate nasal spray (MFNS) twice daily (BID) for 29 days, plus antibiotic. Appropriate antibiotic therapy amoxicillin/clavulanic acid BID.
  Interventions: Drug: MFNS and antibiotic
- Placebo (Placebo Comparator): Matching placebo nasal spray BID for 29 days, plus amoxicillin/clavulanic acid BID
  Interventions: Drug: Matching Placebo nasal spray plus antibiotic

INTERVENTIONS:
Drug: MFNS and antibiotic — MFNS BID for 29 days plus amoxicillin/clavulanic acid BID for 10 days
  Other Names: Group 1: MFNS + Antibiotic
  Arms: MFNS + Antibiotic
Drug: Matching Placebo nasal spray plus antibiotic — Matching placebo nasal spray BID for 29 days plus amoxicillin/clavulanic acid BID for 10 days
  Other Names: Group 2
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Nasonex® (mometasone furoate nasal spray), when used together with an antibiotic, for the relief of symptoms associated with acute bacterial sinusitis. Efficacy will be based on both subjective (assessment of symptom severity by the patient) and objective measurements (computed tomography [CT] imaging of the sinuses).

ELIGIBILITY:
Inclusion Criteria:

* Must be 12 years of age and older, of either sex, and of any race.
* Must weigh at least 40 kg (88 lb).
* Must be willing to give written informed consent and be able to adhere to dose and visit schedules.
* Must have a clinical diagnosis of acute bacterial sinusitis.
* Must be symptomatic at the Screening and Baseline Visits on the basis of subject assessments of major symptoms score.
* Must have radiographic evidence of sinusitis on CT scans taken at Screening.
* Must be in general good health and free of any clinically significant disease (other than sinusitis) that would interfere with the study schedule or procedures, or compromise the subject's safety.
* A subject's clinical laboratory tests (hematology, blood chemistry, and urinalysis), vital signs, and electrocardiogram (ECG) recordings must be within normal limits or clinically acceptable to the investigator/qualified designee. Any test results that are questionable should be referred to the sponsor.
* A female subject of child-bearing potential must have a negative serum pregnancy (beta-hCG) test at Screening. She must agree to use a medically accepted method of contraception throughout the entire study period. Postmenopausal women will be exempted from the use of contraception during the study. Documented absence of menses for at least 1 year will indicate that a female is postmenopausal. If a pre-menarche female subject begins menstruating during the study, a serum pregnancy test must be done at the next visit. A female subject of child-bearing potential who is not currently sexually active must agree to use a medically accepted method of contraception should she become sexually active while participating in the study.

Exclusion Criteria:

* A subject with moderate to severe persistent asthma that requires daily treatment with inhaled steroids, or an exacerbation of asthma within the past 30 days.
* A history of chronic sinusitis (symptoms lasting greater than 3 months) or having undergone sinus or nasal surgery for chronic sinusitis or nasal polyps.
* A history of symptomatic seasonal allergic rhinitis and who, during the study period, is living in or traveling to locations where the allergen to which he/she is allergic is present.
* Subject with glaucoma or a history of posterior subcapsular cataracts.
* Subject with nasal polyps visible upon physical examination, immotile cilia syndrome, immunodeficiency disease, cystic fibrosis, clinically significant cardiovascular (including rheumatic heart disease), pulmonary, renal, hepatic, metabolic, hematological or neurologic disease that in the investigator's judgment might interfere with the evaluation of the therapy, or subjects who are immunocompromised, in renal failure, or on dialysis.
* Subject fails to observe the medication washout times outlined in the protocol prior to Screening.
* Subject has an allergy to corticosteroids or penicillins.
* Subject has used any investigational drug within 30 days of Screening.
* Subject has a concurrent need for antibiotic therapy other than study drug (amoxicillin/clavulanic acid).
* Subject is anticipating sinus or nasal surgery within the next month.
* Subject has been previously randomized into this study.
* Subject is part of the staff personnel directly involved with the study or is a family member of the investigational study staff involved in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Mometasone Furoate Nasal Spray (MFNS): Mometasone furoate nasal spray (MFNS) twice daily (BID) for 29 days, plus antibiotic for 10 days (amoxicillin 875 mg/clavulanic acid 125 mg BID for participants 12 to 15 years of age or amoxicillin 2 gm/clavulanic acid 125 mg BID for participants 16 years of age or older).
- Placebo: Matching placebo nasal spray BID for 29 days, plus antibiotic for 10 days (amoxicillin 875 mg/clavulanic acid 125 mg BID or amoxicillin 2 gm/clavulanic acid 125 mg BID, depending on age).
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Started | 114 | 123
Completed | 98 | 94
Not Completed | 16 | 29
Not completed — Adverse Event | 4 | 6
Not completed — Treatment Failure | 1 | 6
Not completed — Lost to Follow-up | 4 | 7
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Protocol Violation | 1 | 3
Not completed — Did not meet protocol eligibility | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo | Total
Number analyzed (Participants) | 114 | 123 | 237
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 11
  Between 18 and 65 years | 106 | 107 | 213
  >=65 years | 3 | 10 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (13.2) | 39.0 (14.9) | 39.2 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 72 | 152
  Male | 34 | 51 | 85

OUTCOME MEASURES:

1. Primary Outcome: Baseline Change in AM/PM PRIOR Major Symptoms Score (Mss) Minus Sinus Headache Averaged Over Days 1 to 29.
Description: The least squares mean decrease from Baseline in AM/PM PRIOR MSS, excluding sinus headache, averaged over Days 1 to 29. PRIOR is the subject's status over the previous 12 hours (reflective). The MSS was defined as the sum of the following subject-evaluated symptoms: facial pain/pressure/tenderness, sinus headache, purulent rhinorrhea, post-nasal drip, and nasal stuffiness/congestion.MSS scores are as follows: 0=none, 1=mild, 2=moderate, 3=severe for each individual symptom.
Time Frame: 29-day Treatment Period and 2-week no-treatment Follow-up Period.
Population: Not every randomized subject had complete data therefore the number of participants analyzed and the number of participants in the participant flow do not match.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Number analyzed (Participants) | 99 | 103
Units on a scale
  Baseline | 8.57 (1.78) | 8.78 (2.03)
  Days 1-29 | -4.9 (2.69) | -4.46 (2.54)
  Days 30-43 (follow-up) | -6.59 (2.81) | -5.77 (2.98)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray (MFNS) vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.44, 95% CI [-1.14 to 0.25] — For days 1-29
Statistical Analysis 2: Comparison: Mometasone Furoate Nasal Spray (MFNS) vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.82, 95% CI [-1.65 to 0.00] — For follow-up days 30-43

2. Primary Outcome: Change From Baseline to Endpoint in Percent of Opacification of the Maxillary Sinus That Had the Maximum Opacification Score at Baseline
Description: A coronal computerized tomography was obtained to visulaize all nasal sinuses and the ostiomeatal complex. Opacification was measured as a percentage of the area of the sinus that was occupied by either fluid or mucosal thickening. The change in percentage of opacification of one maxillary sinus (the one with the highest percentage of opacification) as compared to antibiotic treatment alone. The percentage of opacification was measured and the change from baseline for that percentage was reported.
Time Frame: 29-day Treatment Period and 2-week no-treatment Follow-up Period.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of opacification
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Number analyzed (Participants) | 99 | 103
Percentage of opacification
  Baseline | 50.7 (30.4) | 56.8 (31.7)
  Change from Baseline at Endpoint | -23.7 (35.2) | -32.5 (32.0)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray (MFNS) vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = 8.8, 95% CI [-0.5 to 18.2] — Change from baseline to endpoint

ADVERSE EVENTS:
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/114 | 1/123
Other Adverse Events (participants affected / at risk) | 22/114 | 17/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate Nasal Spray (MFNS) (N=114) | Placebo (N=123)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate Nasal Spray (MFNS) (N=114) | Placebo (N=123)
Diarrhoea (Gastrointestinal disorders) | 17 (19) | 14 (14)
Fungal Infection (Infections and infestations) | 6 (6) | 3 (4)
Headache (Nervous system disorders) | 6 (7) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to a very high screening failure rate (mainly caused by the necessity to demonstrate CT changes at baseline indicative of acute sinusitis), which limits any conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less